CLINICAL TRIAL: NCT05636306
Title: A Phase 1, Randomized, Placebo Controlled, Double-Blind, Single Dose Escalation Study of NoNO-42 in Healthy Adults
Brief Title: A Phase 1 Study to Evaluate Safety and Tolerability of NoNO-42 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NoNO Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: NoNO42-01
Record Dates: First submitted 2022-11-22; First posted 2022-12-05 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: First-In-Human Study to Evaluate Safety of a New Drug Intended for Treatment of Acute Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NoNO-42 (Experimental): A single intravenous infusion weight-based dose of NoNO-42 administered over 10±1 minute
  Interventions: Drug: NoNO-42
- Placebo (Placebo Comparator): A volume of 0.9% normal saline matching the volume required for a weight-based dosing of NoNO-42, administered as a single 10±1 minute intravenous infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NoNO-42 — A single intravenous infusion weight-based dose of NoNO-42 administered over 10±1 minute
  Arms: NoNO-42
Drug: Placebo — A volume of 0.9% normal saline matching the volume required for a weight-based dosing of NoNO-42, administered as a single 10±1 minute intravenous infusion.
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to evaluate the safety, tolerability and pharmacokinetics of a single ascending intravenous dose of NoNO-42 administered to healthy adults.

Participants will be administered a single intravenous dose of NoNO-42 or placebo.

Participants will be confined for 24 hours post dose with a follow-up visit at Day 4 and Day 28.

DETAILED DESCRIPTION:
The trial was a single, adaptive dose, dose escalation study in healthy male and female adults.

The trial was randomized, double-blind, placebo controlled and evaluated the safety, tolerability, and PK of IV NoNO-42 in healthy adults. Each healthy volunteer was administered a single IV dose of study drug or placebo.

It was planned that up to 10 dosing cohorts would be evaluated. A cohort may have been repeated or added if necessary. Cohort 1 included 4 healthy volunteers (1:1 randomization of NoNO-42 to placebo) with a sentinel dose of 2 healthy volunteers (1:1). Cohorts 2 to 10 were to include 10 new healthy volunteers dosed at each dose level (4:1 randomization of NoNO-42 to placebo) during the single dose escalation. Sentinel dosing with 2 healthy volunteers (1:1) occurred at each dose escalation. Both the dose concentration and the dosing duration may have been adjusted.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures, clinic visits, blood draws, and availability for the duration of the study
* Healthy adult male or female aged 18 to 60 years old.
* Body mass index (BMI) within 18.5 kg/m2 to 30.0 kg/m2, inclusively
* Body weight less than or equal to 120 kg
* Good bilateral venous access sufficient for IV infusions as judged by the investigator or designee
* Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination (including vital signs) and/or ECG, as determined by an investigator

Exclusion Criteria:

* Female who is lactating or pregnant
* History of significant hypersensitivity to NoNO-42 or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
* Presence or history of significant gastrointestinal, liver or kidney disease, or surgery that may affect drug bioavailability
* History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic, renal, hepatic, or dermatologic disease
* Presence of clinically significant ECG abnormalities, or any QT interval abnormalities, at the screening visit, as defined by medical judgment
* Immunization with a COVID-19 vaccine in the 14 days prior to the first study drug administration or plans for vaccination
* Blood pressure below 100 mmHg systolic and 60 mmHg diastolic, and any upper limit is deemed clinically significant by the investigator
* Estimated glomerular filtration rate (eGFR) of <60 mL/min.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Frequency of AEs, abnormal laboratory findings and abnormal vital signs | 28 days
  * Incidence, severity, and causal relationship of AEs.
  * Incidence of abnormal laboratory findings, including histamine.
  * Incidence of abnormal vital signs (blood pressure, heart rate, temperature) and electrocardiogram (ECG) parameters

SECONDARY OUTCOMES:
Pharmacokinetics of NoNO-42 following administration of a single ascending IV dose | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences Company Inc., Mount Royal, Quebec, Canada